CLINICAL TRIAL: NCT06965348
Title: The Acute Effect of Kinesio Taping Applied to the Hamstring and Quadriceps Muscles on Balance and Proprioception in Healthy Young Adult Males: A Randomized Controlled Trial
Brief Title: The Acute Effect of Kinesio Taping on Balance and Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, MİNE PEKESEN KURTÇA, Ass.Prof., Ondokuz Mayıs University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: SÜKAEK-2023 20/15
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-05

CONDITIONS: Healthy Sedanters; Balance; Proprioception
Keywords: Kinesio Taping; Proprioception; Balance; Acute Effect

STUDY DESIGN:
Intervention Model Description: Each participant will receive both the real kinesio taping and placebo taping interventions. One leg will be randomly assigned to the experimental (real taping) condition and the other leg to the control (placebo) condition. This within-subject crossover design allows for direct comparison of intervention effects.
Who Masked: Participant, Outcomes Assessor
Masking Description: In this double-blind study, both the participants and the outcomes assessor were masked to the type of kinesio taping (real or placebo) applied to each leg. The kinesio tape was applied by a separate researcher who did not participate in any of the assessments. Participants were unaware of which leg received the real intervention and which received the placebo taping. This approach was used to minimize bias in both participant response and outcome measurement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application of kinesio tape (Experimental): It will be applied as a facilitating taping technique for the quadriceps and hamstring muscle group as described by Kase et al. The tape will be applied from the muscle origin to its insertion (proximal to distal) for facilitation. The ends of the tape will be rounded to prevent peeling of the tape edges and to increase the length of the tape application.
  For the hamstring muscle group, the application will be applied from the proximal to the distal of the muscle up to the lateral and medial heads of the gastrocnemius muscle. The tape will also be applied to the quadriceps muscle from the proximal to the distal of the muscle, ending on the undersurface of the patella.
  The physiotherapist places the tape base without tension in the first 5 centimeters of the starting point of the hamstring muscles and quadriceps muscle. Light to moderate tension (25-50%) is applied for facilitation. The tail parts of the tape are placed on the skin without tension at a distance of 2 to 5 cm from the e
  Interventions: Device: Application of kinesio tape
- Control group (Placebo Comparator): For the quadriceps and hamstring muscle group, kinesio tape will be applied from the muscle origin to the insertion (proximal to distal) without any tension. The ends of the tape will be rounded to prevent peeling of the tape edges and to increase the length of the tape application.
  For the hamstring muscle group, the application will be applied from the proximal to the distal of the muscle up to the lateral and medial heads of the gastrocnemius muscle. The tape will also be applied to the quadriceps muscle from the proximal to the distal of the muscle, ending at the lower surface of the patella.
  Interventions: Other: Placebo Group

INTERVENTIONS:
Device: Application of kinesio tape — The facilitating taping technique for the quadriceps and hamstring muscle group described by Kase et al. will be applied to the kinesio tape group. The tape will be applied from the muscle origin to the insertion (proximal to distal) for facilitation.
  The application for the hamstring muscle group will be applied from the proximal to the distal of the muscle up to the lateral and medial heads of the gastrocnemius muscle. The tape will be applied to the quadriceps muscle from the proximal to the distal of the muscle, ending on the undersurface of the patella.
  The physiotherapist places the tape base without tension in the first 5 centimeters of the starting point of the hamstring muscles and quadriceps muscle. Light to moderate tension (25-50%) is applied for facilitation. The tail parts of the tape are placed on the skin without tension at a distance of 2 to 5.
  Arms: Application of kinesio tape
Other: Placebo Group — The application for the hamstring muscle group will be applied from the proximal to the distal of the muscle up to the lateral and medial heads of the gastrocnemius muscle. The tape will also be applied to the quadriceps muscle from the proximal to the distal of the muscle, ending at the lower surface of the patella.The placebo group will have tape applied to the quadriceps and hamstring muscle groups without any tension.
  Arms: Control group

SUMMARY:
Kinesio tape will be applied to the leg muscles of two groups of healthy and young participants using a specific taping technique. After the application of the tape, assessments of balance and proprioception will be conducted. The taping will be performed bilaterally on both legs, and for all participants, taped and untaped measurements will be carried out bilaterally on alternating days within the same week.

Prior to the assessments, all participants will be asked to complete a 5-minute warm-up session on a bicycle ergometer, followed by four sets of 30-second static stretching exercises for the leg and hip muscles, with 30-second rest intervals between each set.

In this way, the acute effects of kinesio taping on balance and proprioception will be investigated.

DETAILED DESCRIPTION:
This study aims to examine the acute effects of kinesio taping (KT) applied to the hamstring and quadriceps muscle groups on balance and proprioception in healthy young male individuals.

The primary objective of the study is to determine whether kinesio taping enhances proprioceptive feedback in the targeted muscle groups and whether this has a short-term impact on postural balance. As balance and proprioception are critically important for daily functional activities and sports performance, they will be evaluated using objective assessment methods in this research.

The study will include 20 healthy and voluntary male participants. Participants will be divided into two groups: real taping and placebo taping. For each participant, one leg will be randomly assigned to the experimental group (real KT application), and the other leg to the control group (placebo). All interventions and assessments will be conducted in a double-blind design, where the assessor will not know which leg received which application.

All participants will begin with a 5-minute warm-up on a bicycle ergometer, followed by four sets of 30-second static stretching exercises targeting the hamstring, quadriceps, and gluteal muscles, with 30-second rest intervals between sets. The kinesio tape will be applied using the facilitation technique described by Kase et al., from origin to insertion (proximal to distal).

Proprioception will be assessed using an isokinetic dynamometer through the Active Joint Position Reproduction (AJPR) test. Participants will be asked to actively reproduce specific knee angles, and the differences between the actual and reproduced angles will be recorded for analysis.

Postural balance will be assessed using the CSMI-TecnoBody PK-252 balance analysis system, through both static and dynamic tests. In the static test, participants will stand on a stable platform with eyes open while their balance is measured. In the dynamic test, participants will follow a predefined movement path using their feet on a moving platform to assess balance performance.

At the end of the study, the collected data will be statistically analyzed to determine whether kinesio taping has an acute positive effect on balance and proprioception. The findings will be evaluated for their potential contributions to physical activity, athlete health, and rehabilitation practices.

ELIGIBILITY:
Inclusion Criteria:

Male individuals aged between 18 and 30 years

Healthy with no known musculoskeletal disorders

Voluntarily agrees to participate in the study

Has no contraindications to physical activity or kinesio taping

Provides written informed consent

Exclusion Criteria:

History of musculoskeletal injury within the last 6 months

Presence of any vestibular or auditory disorders

Active cellulitis or skin infection at the application site

Open wounds or history of deep vein thrombosis (DVT)

Known allergy to kinesio tape or related materials

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Joint Position Sense (Proprioception) Measured by Active Joint Position Reproduction Test | Within 30 minutes after kinesio taping application
  Proprioception will be assessed using the Active Joint Position Reproduction (AJPR) test with an isokinetic dynamometer. Participants will be asked to actively replicate three target knee flexion angles after passive teaching. The absolute error between the target angle and the angle reproduced by the participant will be recorded. Three trials will be performed for each angle, and the mean absolute error will be calculated for analysis. A lower error score indicates better proprioceptive accuracy.
Postural Balance Assessment | 3 months
  Before measurements are taken for static and dynamic balance, participants will complete a 10-minute warm-up exercise consisting of 5 minutes of low-intensity running and warm-up exercises. All participants will be allowed to do one trial before the test begins. Then, athletes will be placed on a platform and subjected to open-eye static balance tests. Measurements will be taken with the patient's feet shoulder-width apart on the CSMI-TecnoBody PK-252 balance device platform and the feet on the lines representing the x and y axes of the platform and equidistant from the starting point. The tests will last 30 seconds, the body position will be maintained and the subject's position will be monitored on the screen. The test will be automatically saved at the end of 30 seconds. For Dynamic Balance, subjects will be instructed to complete the test using only the feet to minimize upper body movements.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)